CLINICAL TRIAL: NCT01412866
Title: Electronic Decision Support Systems for Smokers With Severe Mental Illness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: U.S. Department of Education (U.S. Federal Agency); Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Mary F. Brunette, MD, MD, Dartmouth-Hitchcock Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EDSS1
Record Dates: First submitted 2011-08-04; First posted 2011-08-09 (Estimated); Results first posted 2018-12-12 (Actual); Last update posted 2018-12-12 (Actual); Status verified 2018-12

CONDITIONS: Severe Mental Illness; Nicotine Dependence; Schizophrenia; Tobacco Use Disorder
Keywords: schizophrenia; severe mental illness; nicotine; smoking; motivation; electronic decision support system; motivational interviewing
MeSH Terms: conditions — Mental Disorders; Tobacco Use Disorder; Schizophrenia; Smoking

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- EDSS with CO monitor (Experimental): Web-based electronic decision support system (EDSS) with carbon monoxide (CO) monitor and health-checklist
  Interventions: Behavioral: EDSS with CO feedback and health checklist
- EDSS without CO monitor (Active Comparator): Web-based electronic decision support system (EDSS) with health-checklist only
  Interventions: Behavioral: EDSS with health checklist feedback alon

INTERVENTIONS:
Behavioral: EDSS with CO feedback and health checklist — Web-based electronic decision support system with CO feedback and health-checklist
  Arms: EDSS with CO monitor
Behavioral: EDSS with health checklist feedback alon — Web-based electronic decision support system (EDSS) with health-checklist feedback alone (without CO feedback)
  Arms: EDSS without CO monitor

SUMMARY:
This randomized clinical trial among SMI smokers assessed whether the EDSS with carbon monoxide monitor and health-checklist feedback lead to higher rates of initiation of smoking cessation treatment, days of smoking abstinence and Fagerstrom Dependence scores, compared to use of the EDSS with checklist feedback alone.

DETAILED DESCRIPTION:
Up to 80% of Americans with serious mental illnesses (SMI; schizophrenia and severe mood disorders) smoke cigarettes, and most suffer related health consequences. Although combined treatment with medication and psychosocial therapy can help people with SMI to quit smoking, it is rarely used. Motivational interventions can enhance the use of combined treatment, but motivational interventions are expensive and unavailable. To fill this gap, Dartmouth and Thresholds investigators have developed an easy-to-use, web-based electronic decision support system (EDSS) that aims to educate and motivate smokers with SMI. Preliminary testing has demonstrated excellent usability and increased engagement in smoking cessation treatments.

One critical issue is the use of personalized health feedback. Motivational interventions for smoking cessation for smokers with SMI, including our EDSS, have included personal feedback from a breath monitor that measures carbon monoxide, a toxic component of cigarette smoke. Feedback regarding carbon monoxide is thought to motivate the user by personalizing the health risks of smoking. The carbon monoxide monitor is, however, expensive, difficult to implement, and largely unavailable in public mental health and primary care clinics. Further, research on use of carbon monoxide monitoring in the general population is equivocal. Another motivational strategy to personalize the negative health effects of smoking is a health checklist with feedback. Health checklists have been shown to be effective, are easy to use, have no expense, but have not been assessed separately from carbon monoxide monitor feedback among SMI smokers. Testing the effect of feedback from the health checklist compared to feedback from the carbon monoxide monitor is an essential next step in the development of this tool.

Aim 1. The investigators propose a randomized clinical trial among SMI smokers to assess whether the EDSS with carbon monoxide monitor and health-checklist feedback will lead to higher rates of initiation of smoking cessation treatment than the EDSS with health-checklist feedback alone.

Aim 1.a. To explore whether use of the EDSS with carbon monoxide monitor and health-checklist feedback leads to higher rates of the distal outcomes, days of smoking abstinence and Fagerstrom Dependence scores, than use of the EDSS with checklist feedback alone.

ELIGIBILITY:
Inclusion Criteria:

* adult age 18-75
* in treatment for severe mental illness,
* current smoker,
* physically able to use a computer

Exclusion Criteria:

* Using smoking cessation treatment in past month,
* substance dependence with current use

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2011-05; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary F Brunette, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Thresholds Psychiatric Rehabilitation Center, Chicago, Illinois, United States

REFERENCES:
- [Background] Brunette MF, Ferron JC, McHugo GJ, Davis KE, Devitt TS, Wilkness SM, Drake RE. An electronic decision support system to motivate people with severe mental illnesses to quit smoking. Psychiatr Serv. 2011 Apr;62(4):360-6. doi: 10.1176/ps.62.4.pss6204_0360. PMID 21459986
- [Derived] Ferron JC, Devitt T, McHugo GJ, A Jonikas J, Cook JA, Brunette MF. Abstinence and Use of Community-Based Cessation Treatment After a Motivational Intervention Among smokers with Severe Mental Illness. Community Ment Health J. 2016 May;52(4):446-56. doi: 10.1007/s10597-016-9998-1. Epub 2016 Mar 1. PMID 26932324

RESULTS

PARTICIPANT FLOW:
Groups:
- EDSS With CO Monitor Feedback: Electronic decision support system with carbon monoxide (CO) monitor feedback: Web-based electronic decision support system (EDSS) with carbon monoxide monitor and health-checklist
- EDSS Without CO Monitor Feedback: Electronic decision support system without carbon monoxide (CO) monitor feedback: Web-based electronic decision support system (EDSS) with health-checklist feedback alone
Period: Overall Study
Arm/Group | EDSS With CO Monitor Feedback | EDSS Without CO Monitor Feedback
Started | 58 | 66
Completed | 57 | 64
Not Completed | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- EDSS With CO Monitor Feedback: Electronic decision support system with CO monitor feedback: Web-based electronic decision support system (EDSS) with carbon monoxide monitor and health-checklist
- EDSS Without CO Monitor Feedback: Electronic decision support system without CO monitor feedback: Web-based electronic decision support system (EDSS) with health-checklist feedback alone
- Total: Total of all reporting groups
Arm/Group | EDSS With CO Monitor Feedback | EDSS Without CO Monitor Feedback | Total
Number analyzed (Participants) | 58 | 66 | 124
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.7 (9.3) | 46.3 (10.8) | 46.5 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 21 | 35
  Male | 44 | 45 | 89
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American | 30 | 30 | 60
  Caucasian | 26 | 16 | 42
  Hispanic | 6 | 12 | 18
Cigarettes smoked per day [Mean (Standard Deviation); unit: Cigarettes] | 15.0 (11.8) | 15.1 (10.8) | 15.0 (11.2)

OUTCOME MEASURES:

1. Primary Outcome: Initiation of Smoking Cessation Treatment
Description: Started smoking cessation treatment
Time Frame: 2 months
Measure: Number; unit: participants
Arm/Group | EDSS With CO Monitor Feedback | EDSS Without CO Monitor Feedback
Number analyzed (Participants) | 58 | 66
participants | 14 | 24
Statistical Analysis 1: Comparison: EDSS With CO Monitor Feedback vs EDSS Without CO Monitor Feedback; Test type: Superiority or Other; p = 0.08, Chi-squared; df=1

2. Secondary Outcome: Days of Nicotine Abstinence
Time Frame: 6 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | EDSS With CO Monitor Feedback | EDSS Without CO Monitor Feedback
Serious Adverse Events (participants affected / at risk) | 0/58 | 0/66
Other Adverse Events (participants affected / at risk) | 0/58 | 0/66

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No